CLINICAL TRIAL: NCT01701401
Title: A Phase 3, Multicenter, Randomized, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/GS-5885 Fixed-Dose Combination (FDC) +/- Ribavirin for 12 and 24 Weeks in Treatment-Naive Subjects With Chronic Genotype 1 HCV Infection.
Brief Title: Safety and Efficacy of Ledipasvir/Sofosbuvir Fixed-Dose Combination (FDC) With and Without Ribavirin for the Treatment of HCV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-0102; 2012-003387-43 (EudraCT Number)
Record Dates: First submitted 2012-10-02; First posted 2012-10-05 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2015-03

CONDITIONS: Chronic Hepatitis C Virus
Keywords: HCV genotype 1 (GT-1); HCV; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; GS-7977; GS-5885; Ribavirin; Open Label; Sofosbuvir; Additional relevant MeSH terms:; Hepatitis; Hepatitis, Chronic; Hepatitis C; Hepatitis C, Chronic; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Virus Diseases; Enterovirus Infections; Picornaviridae Infections; RNA Virus Infections; Flaviviridae Infections; Antiviral Agents; Anti-Infective Agents; Therapeutic Uses; Pharmacologic Actions; Antimetabolites; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis; Hepatitis, Chronic; Hepatitis C; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Virus Diseases; Enterovirus Infections; Picornaviridae Infections; RNA Virus Infections; Flaviviridae Infections | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LDV/SOF 12 weeks (Experimental): LDV/SOF administered for 12 weeks
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV 12 weeks (Experimental): LDV/SOF+RBV administered for 12 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV
- LDV/SOF 24 weeks (Experimental): LDV/SOF administered for 24 weeks
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV 24 weeks (Experimental): LDV/SOF+RBV administered for 24 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV

INTERVENTIONS:
Drug: LDV/SOF — LDV/SOF 90/400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
Drug: RBV — RBV tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: LDV/SOF+RBV 12 weeks; LDV/SOF+RBV 24 weeks

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and antiviral efficacy of ledipasvir (LDV)/sofosbuvir (SOF) fixed-dose combination (FDC) tablets with or without ribavirin (RBV) administered for 12 and 24 weeks in treatment-naive subjects with chronic genotype 1 HCV infection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, with chronic genotype 1 HCV infection
* HCV treatment-naive
* HCV RNA > 10,000 IU/mL at screening
* Cirrhosis determination; a liver biopsy may be required
* Screening laboratory values within defined thresholds
* Use of two effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Co-infection with HIV or hepatitis B virus (HBV)
* Current or prior history of clinical hepatic decompensation
* Hepatocellular carcinoma (HCC) or other malignancy (with exception of certain resolved skin cancers)
* Chronic use of systemic immunosuppressive agents
* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Yang, Pharm D, Study Director — Gilead Sciences
Locations (88):
- United States (53):
  - Birmingham, Alabama
  - La Jolla, California
  - Long Beach, California
  - Los Angeles, California
  - Palo Alto, California
  - Sacramento, California
  - San Diego, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Lutherville, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Rochester, Minnesota
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Hillsborough, New Jersey
  - Albuquerque, New Mexico
  - Santa Fe, New Mexico
  - Manhasset, New York
  - New York, New York
  - The Bronx, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Fayetteville, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Fairfax, Virginia
  - Falls Church, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
- France (8):
  - CHRU Lille
  - Clichy
  - Créteil
  - La Tronche
  - Lyon
  - Marseille
  - Nice
  - Paris
- Germany (9):
  - Berlin
  - Cologne
  - Düsseldorf
  - Essen
  - Frankfurt
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - Mainz
- Italy (8):
  - Bologna
  - Brescia
  - Milan
  - Padua
  - Palermo
  - Roma
  - San Giovanni Rotondo
  - Torino
- San Juan, Puerto Rico
- Spain (5):
  - Barcelona
  - Madrid
  - Málaga
  - Santander
  - Seville
- United Kingdom (4):
  - Birmingham, Wstmid
  - London
  - Manchester
  - Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] Grebely J, Mauss S, Brown A, Bronowicki JP, Puoti M, Wyles D, Natha M, Zhu Y, Yang J, Kreter B, Brainard DM, Yun C, Carr V, Dore GJ. Efficacy and Safety of Ledipasvir/Sofosbuvir With and Without Ribavirin in Patients With Chronic HCV Genotype 1 Infection Receiving Opioid Substitution Therapy: Analysis of Phase 3 ION Trials. Clin Infect Dis. 2016 Dec 1;63(11):1405-1411. doi: 10.1093/cid/ciw580. Epub 2016 Aug 23. PMID 27553375
- [Derived] Younossi ZM, Elsheikh E, Stepanova M, Gerber L, Nader F, Stamm LM, Brainard DM, McHutchinson JG. Ledipasvir/sofosbuvir treatment of hepatitis C virus is associated with reduction in serum apolipoprotein levels. J Viral Hepat. 2015 Dec;22(12):977-82. doi: 10.1111/jvh.12448. Epub 2015 Aug 17. PMID 26280786
- [Derived] Afdhal N, Zeuzem S, Kwo P, Chojkier M, Gitlin N, Puoti M, Romero-Gomez M, Zarski JP, Agarwal K, Buggisch P, Foster GR, Brau N, Buti M, Jacobson IM, Subramanian GM, Ding X, Mo H, Yang JC, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Mangia A, Marcellin P; ION-1 Investigators. Ledipasvir and sofosbuvir for untreated HCV genotype 1 infection. N Engl J Med. 2014 May 15;370(20):1889-98. doi: 10.1056/NEJMoa1402454. Epub 2014 Apr 11. PMID 24725239

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 100 study sites in the United States and Europe. The first participant was screened on 26 September 2012. The last study visit occurred on 30 April 2014.
Pre-assignment Details: 1015 participants were screened.
Groups:
- LDV/SOF 12 Weeks: Ledipasvir/sofosbuvir (LDV/SOF) 90/400 mg FDC tablet once daily for 12 weeks
- LDV/SOF+RBV 12 Weeks: LDV/SOF 90/400 mg FDC tablet once daily plus ribavirin (RBV) tablets (1000 to 1200 mg daily based on weight) in a divided daily dose for 12 weeks
- LDV/SOF 24 Weeks: LDV/SOF 90/400 mg FDC tablet once daily for 24 weeks
- LDV/SOF+RBV 24 Weeks: LDV/SOF 90/400 mg FDC tablet once daily plus RBV tablets (1000 to 1200 mg daily based on weight) in a divided daily dose for 24 weeks
Period: Overall Study
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Started | 217 | 218 | 217 | 218
Completed | 207 | 209 | 212 | 212
Not Completed | 10 | 9 | 5 | 6
Not completed — Randomized But Not Treated | 3 | 1 | 0 | 1
Not completed — Lost to Follow-up | 5 | 5 | 1 | 3
Not completed — Withdrew Consent | 0 | 3 | 1 | 2
Not completed — Lack of Efficacy | 1 | 0 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants were randomized and received at least 1 dose of study drug.
Groups:
- LDV/SOF 12 Weeks: LDV/SOF 90/400 mg FDC tablet once daily for 12 weeks
- LDV/SOF+RBV 12 Weeks: LDV/SOF 90/400 mg FDC tablet once daily plus RBV tablets (1000 to 1200 mg daily based on weight) in a divided daily dose for 12 weeks
- Total: Total of all reporting groups
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks | Total
Number analyzed (Participants) | 214 | 217 | 217 | 217 | 865
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (10.7) | 52 (11.5) | 53 (10.3) | 53 (9.9) | 52 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 89 | 78 | 98 | 352
  Male | 127 | 128 | 139 | 119 | 513
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 24 | 26 | 32 | 26 | 108
  White | 187 | 188 | 177 | 183 | 735
  Asian | 1 | 0 | 5 | 5 | 11
  American Indian/Alaska Native | 0 | 1 | 0 | 1 | 2
  Hawaiian or Pacific Islander | 0 | 0 | 1 | 0 | 1
  Other | 2 | 1 | 2 | 1 | 6
  Not Disclosed | 0 | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 26 | 20 | 29 | 26 | 101
  Not Hispanic or Latino | 187 | 197 | 188 | 190 | 762
  Not Disclosed | 1 | 0 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  France | 11 | 24 | 18 | 10 | 63
  United States | 125 | 118 | 132 | 137 | 512
  Spain | 14 | 15 | 12 | 14 | 55
  Germany | 24 | 20 | 22 | 18 | 84
  United Kingdom | 13 | 17 | 10 | 15 | 55
  Italy | 27 | 23 | 23 | 23 | 96
Hepatitis C Virus (HCV) RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.4 (0.69) | 6.4 (0.64) | 6.3 (0.68) | 6.3 (0.65) | 6.4 (0.66)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 45 | 44 | 49 | 44 | 182
  ≥ 800,000 IU/mL | 169 | 173 | 168 | 173 | 683
HCV Genotype [Number; unit: participants] — There are variations of HCV which are all similar enough to be called HCV, but are distinct enough to be referred to as HCV genotypes.
  participants
    Genotype 1a | 144 | 148 | 146 | 143 | 581
    Genotype 1b | 66 | 68 | 68 | 71 | 273
    Genotype 1 (no confirmed subtype) | 1 | 1 | 1 | 1 | 4
    Genotype 4 | 1 | 0 | 0 | 1 | 2
    Missing | 2 | 0 | 2 | 1 | 5
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 55 | 76 | 52 | 73 | 256
    CT | 113 | 107 | 119 | 112 | 451
    TT | 46 | 34 | 46 | 32 | 158

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Study Drug (SVR12)
Description: SVR12 was defined as HCV RNA level < the lower limit of quantification (LLOQ, ie, < 25 copies/mL) 12 weeks after last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 214 | 217 | 217 | 217
percentage of participants | 98.6 | 97.2 | 98.2 | 99.1
Statistical Analysis 1: Comparison: LDV/SOF 12 Weeks; Test type: Superiority or Other; p < 0.001, Binomial test — The p-value for the comparison of the LDV/SOF 12 week group against the adjusted historical null rate (60%) was based on a 2-sided 1-sample binomial test
Statistical Analysis 2: Comparison: LDV/SOF+RBV 12 Weeks; Test type: Superiority or Other; p < 0.001, Binomial test — The p-value for the comparison of the LDV/SOF+RBV 12 week group against the adjusted historical null rate (60%) was based on a 2-sided 1-sample binomial test
Statistical Analysis 3: Comparison: LDV/SOF 24 Weeks; Test type: Superiority or Other; p < 0.001, Binomial test — The p-value for the comparison of the LDV/SOF 24 week group against the adjusted historical null rate (60%) was based on a 2-sided 1-sample binomial test
Statistical Analysis 4: Comparison: LDV/SOF+RBV 24 Weeks; Test type: Superiority or Other; p < 0.001, Binomial test — The p-value for the comparison of the LDV/SOF+RBV 24 week group against the adjusted historical null rate (60%) was based on a 2-sided 1-sample binomial test

2. Primary Outcome: Incidence of Adverse Events Leading to Permanent Discontinuation From Any Study Drug
Description: The percentage of participants who experienced an adverse event leading to permanent discontinuation from any study drug was summarized.
Time Frame: Up to 24 weeks
Population: Safety Analysis Set: participants were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 214 | 217 | 217 | 217
percentage of participants | 0 | 0.5 | 1.8 | 3.7

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Study Drug
Description: SVR4 and SVR24 were defined as HCV RNA level < LLOQ at 4 and 24 weeks after discontinuation of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 214 | 217 | 217 | 217
percentage of participants
  SVR4 | 98.6 | 98.2 | 99.1 | 99.1
  SVR24 | 98.6 | 97.2 | 98.2 | 99.1

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 2
Time Frame: Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 213 | 217 | 216 | 217
percentage of participants | 82.2 | 83.4 | 82.9 | 82.9

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 4
Time Frame: Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 213 | 217 | 216 | 217
percentage of participants | 100 | 99.1 | 100 | 100

6. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 8
Time Frame: Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 213 | 215 | 215 | 217
percentage of participants | 99.5 | 100 | 99.5 | 100

7. Secondary Outcome: Change From Baseline in HCV RNA at Week 2
Time Frame: Baseline; Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 213 | 217 | 216 | 216
log10 IU/mL | -4.90 (0.657) | -4.94 (0.633) | -4.86 (0.670) | -4.89 (0.648)

8. Secondary Outcome: Change From Baseline in HCV RNA at Week 4
Time Frame: Baseline; Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 213 | 216 | 216 | 217
log10 IU/mL | -4.99 (0.697) | -5.02 (0.623) | -4.93 (0.678) | -4.96 (0.651)

9. Secondary Outcome: Change From Baseline in HCV RNA at Week 8
Time Frame: Baseline; Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 213 | 215 | 216 | 217
log10 IU/mL | -4.99 (0.696) | -5.02 (0.625) | -4.91 (0.702) | -4.96 (0.651)

10. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: On-treatment virologic failure was defined as:
  * Breakthrough: HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ, while on treatment, confirmed with 2 consecutive values (second confirmation value could have been posttreatment), or last available on-treatment measurement with no subsequent follow- up values, OR
  * Rebound: > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment, confirmed with 2 consecutive values (second confirmation value could have been posttreatment), or last available on-treatment measurement with no subsequent follow-up values, OR
  * Nonresponse: HCV RNA persistently ≥ LLOQ through 8 weeks of treatment
  Virologic relapse was defined as HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement
Time Frame: Baseline to posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 214 | 217 | 217 | 217
percentage of participants
  On-treatment virologic failure | 0 | 0 | 0.5 | 0
  Virologic relapse | 0.5 | 0 | 0.5 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set: participants were randomized and received at least 1 dose of study drug.
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Serious Adverse Events (participants affected / at risk) | 1/214 | 7/217 | 18/217 | 7/217
Other Adverse Events (participants affected / at risk) | 140/214 | 168/217 | 149/217 | 189/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks (N=214) | LDV/SOF+RBV 12 Weeks (N=217) | LDV/SOF 24 Weeks (N=217) | LDV/SOF+RBV 24 Weeks (N=217)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Factor VIII inhibition (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 0 | 1 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Substance abuse (Psychiatric disorders) | 0 | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks (N=214) | LDV/SOF+RBV 12 Weeks (N=217) | LDV/SOF 24 Weeks (N=217) | LDV/SOF+RBV 24 Weeks (N=217)
Anaemia (Blood and lymphatic system disorders) | 0 | 25 | 0 | 22
Nausea (Gastrointestinal disorders) | 24 | 37 | 29 | 32
Diarrhoea (Gastrointestinal disorders) | 24 | 18 | 24 | 14
Constipation (Gastrointestinal disorders) | 13 | 12 | 15 | 10
Dyspepsia (Gastrointestinal disorders) | 7 | 11 | 14 | 12
Abdominal pain (Gastrointestinal disorders) | 12 | 9 | 7 | 8
Vomiting (Gastrointestinal disorders) | 7 | 9 | 6 | 12
Abdominal pain upper (Gastrointestinal disorders) | 5 | 11 | 7 | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 7 | 3 | 11
Fatigue (General disorders) | 46 | 79 | 53 | 84
Asthenia (General disorders) | 14 | 23 | 20 | 26
Irritability (General disorders) | 11 | 17 | 17 | 24
Nasopharyngitis (Infections and infestations) | 14 | 9 | 13 | 19
Decreased appetite (Metabolism and nutrition disorders) | 10 | 12 | 8 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 14 | 21 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 13 | 12 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 5 | 12 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 14 | 9 | 12
Headache (Nervous system disorders) | 54 | 50 | 54 | 66
Dizziness (Nervous system disorders) | 11 | 10 | 14 | 18
Insomnia (Psychiatric disorders) | 17 | 45 | 26 | 46
Anxiety (Psychiatric disorders) | 7 | 9 | 12 | 19
Depression (Psychiatric disorders) | 5 | 6 | 5 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 22 | 16 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 18 | 5 | 15
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 9 | 2 | 11
Rash (Skin and subcutaneous tissue disorders) | 16 | 21 | 16 | 26
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 22 | 8 | 20
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 14 | 3 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years